CLINICAL TRIAL: NCT03161938
Title: High vs Low Dose Dexamethasone on Complications in the Immediate Postoperative Phase After Periacetabular (GANZ) Osteotomy
Brief Title: High vs Low Dose Dexamethasone on Complications in the Immediate Postoperative Phase
Acronym: DEX-GANZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristin Julia Steinthorsdottir, MD, clinical assistant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEXGANZ01
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Hip Dysplasia; Postoperative Complications
MeSH Terms: conditions — Hip Dislocation; Postoperative Complications | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone 48 mg (Active Comparator): Dexamethasone 48 mg pre-operative, single shot injection
  Interventions: Drug: Dexamethasone
- Dexamethasone 8 mg (Active Comparator): Dexamethasone 8 mg pre-operative, single shot injection
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — intravenous

SUMMARY:
The aim of this study is to investigate the effect of a single preoperative high-dose steroid injection on complications in the immediate postoperative phase after periacetabular osteotomy. Primary outcome is the proportion of patients who have moderate to severe postoperative pain in the post anaesthesia care unit. Secondary outcomes are organspecific complications in the post anaesthesia phase, pain and nausea the first 5 days, wound infection and readmissions the first 30 days after surgery.

The investigators hypothesize that the frequency of moderate to severe pain and organspecific complications in the post anaesthesia care unit will be lower among patients receiving high dose dexamethasone. The investigators hypothesize, that there will be no difference in wound infections or readmissions.

DETAILED DESCRIPTION:
Post-surgery, patients are traditionally observed and treated in post-anesthesia care units (PACU) until they are discharged to the ward (or directly home) assessed by standardized international discharge criteria.

The research project "Why in PACU?" (Rigshospitalet, Denmark), has since the beginning of 2016 systematically collected and analyzed procedure-related complications in the recovery phase. The complications include pain, nausea/vomiting, circulatory and respiratory problems, orthostatic intolerance and cognitive disorders. Common to all the above-mentioned post-operative problems are the possible links to the inflammatory response caused by the surgical trauma.

Glucocorticoids can in this context be central for the reduction of acute postoperative organ dysfunctions, caused by the anti-inflammatory effect. In a number of different surgical procedures, single dose, pre-operative glucocorticoids have been shown to reduce post-operative nausea and vomiting (PONV), acute pain and need of opioids as well as accelerate the convalescence.

Meta-analyses also showed that single-dose administration of glucocorticoids (methylprednisolone and dexamethasone) for surgical patients is safe as opposed to long-term treatment.

The "Why in PACU?" database shows that 70 % of patients experience moderate to severe pain in the immediate postoperative phase. This is despite a multimodal analgesic regime with preoperative analgesics and local analgesic catheter in the surgical site.

Opioids are frequently administered to relieve pain, resulting in sedation, risk of hypoxia and delaying mobilization.

Patients having Ganz osteotomy are primarily young women with hipdysplasia, that are otherwise healthy. Lenght of stay is typically 5 days, due to pain and lack of mobilisation.

In this study patients are randomized to either high dose (48 mg) or standard/low dose (8 mg) dexamethasone, administered preoperatively. The hypothese is that patients receiving high dose dexamethasone will experience less pain in the immediate postoperative course and receive less opioids.

The study is not placebo-controlled since the positive effects of dexamethasone 8 mg on PONV have been shown in numerous trials, and is already being administered to all patients at the clinic. It would therefore not be ethically correct to withdraw from this practise.

ELIGIBILITY:
Inclusion Criteria:

* planned unilateral periacetabular osteotomy
* informed signed consent

Exclusion Criteria:

* Chronic/ongoing (<30 days) use of glucocorticoids (except inhalation therapy)
* ongoing (<30 days) use of immunosuppressive therapy
* insulin dependent diabetes
* pregnancy/breastfeeding
* allergies toward study medication, or medication in the standard treatment
* surgery cannot be performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: kristin J Steinthorsdottir, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steinthorsdottir KJ, Awada HN, Dirks J, Sturup J, Winther NS, Kehlet H, Aasvang EK. Early postoperative recovery after peri-acetabular osteotomy: A double-blind, randomised single-centre trial of 48 vs. 8 mg dexamethasone. Eur J Anaesthesiol. 2021 Mar 1;38(Suppl 1):S41-S49. doi: 10.1097/EJA.0000000000001410. PMID 33399374

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (8) | 29 (7) | 29 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 5 | 8 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23 (3) | 23 (3) | 23 (3)
Previous operation (contralateral periacetabular osteotomy) [Count of Participants; unit: Participants] | 3 | 9 | 12
Comorbidities, none [Count of Participants; unit: Participants] | 30 | 27 | 57
Daily intake of analgesics, preoperative [Count of Participants; unit: Participants] | 4 | 6 | 10
Daily intake of opioids, preoperative [Count of Participants; unit: Participants] | 2 | 2 | 4
Operating time [Mean (Standard Deviation); unit: minutes] | 71 (20) | 69 (13) | 70 (17)
Bleeding [Mean (Standard Deviation); unit: ml] | 467 (301) | 510 (295) | 500 (296)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Moderate to Severe Postoperative Pain
Description: Moderate to severe pain (NRS > 3) in the post-anesthesia care unit (PACU)
Time Frame: 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 32 | 32
Participants | 26 | 22
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Null hypothesis: Patients receiving 48 mg of preoperative dexamethasone have less postoperative pain. Power calculation: Acute pain is reduced from 70% to 35% for patients receiving 48 mg of dexamathesone, 80% power, 0.05 statistical significance level; Test type: Superiority; p = 0.248, Chi-squared, Corrected; Odds Ratio (OR) = 0.508, 95% CI 2-sided [0.159 to 1.620]

2. Secondary Outcome: Lenght of Stay, PACU
Description: Total lenght of stay in PACU
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 32 | 32
hours | 2 [2 to 3] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Test type: Superiority; p = 0.519, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Lenght of Stay, Hospital
Description: Total lenght of stay, Hospital
Time Frame: 1 week
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 32 | 32
hours | 78 [73 to 101] | 77 [71 to 94]
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Test type: Superiority; p = 0.468, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Pain Scores, PACU
Description: Differences between groups in maximal and average pain score during PACU stay. Pain scores are measured on a numeric rating scale (NRS), 0-10. 0 is no pain, 10 is worst pain imaginable.
Time Frame: 12 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale (numeric rating scale)
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 32 | 32
score on a scale (numeric rating scale)
  Maximal pain | 5 [3 to 7] | 5 [3 to 7]
  Average pain | 2 [1 to 3] | 2 [1 to 3]
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Maximal pain; Test type: Superiority; p = 0.913, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Average pain; Test type: Superiority; p = 0.722, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Complications
Description: Patients with complications requiring treatment the first 24 hours (PACU and ward)
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 32 | 32
Participants | 24 | 25
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Test type: Superiority; p = 0.768, Chi-squared, Corrected; Odds Ratio (OR) = 1.190, 95% CI 2-sided [0.374 to 3.793]

6. Secondary Outcome: Self Reported Postoperative Pain
Description: Self-reported pain on a Numeric rating scale (NRS), NRS 0-10, 0 = no pain, 10= worst pain imaginable.
  Reported once daily, postoperative days 0 to 4
Time Frame: postoperative day 0 to 4, once a day
Population: Missing data, missing at random
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 26 | 25
score on a scale
  Day 0 | 3 (2) | 4 (2)
  Day 1 | 4 (2) | 4 (2)
  Day 2 | 3 (2) | 4 (2)
  Day 3: number analyzed (Participants) | 24 | 23
  Day 3 | 3 (2) | 3 (2)
  Day 4: number analyzed (Participants) | 22 | 20
  Day 4 | 3 (2) | 3 (2)
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Test type: Superiority; p = 0.133, Regression, Linear

7. Secondary Outcome: Number of Patients With Post Operative Nausea and Vomiting (PONV) Postoperative Days 0 to 4
Description: Patients reporting PONV and/or receiving antiemetic medication on postoperative days 0 to 4
Time Frame: postoperative day 0 to 4, once a day
Population: Missing data day 4 due to discharge from hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 32 | 32
Participants
  Day 0 | 7 | 8
  Day 1 | 6 | 9
  Day 2 | 9 | 11
  Day 3 | 7 | 4
  Day 4: number analyzed (Participants) | 23 | 24
  Day 4 | 3 | 2
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 0; Test type: Superiority; p = 0.768, Chi-squared, Corrected — Not adjusted for multiple comparisons, statistical level of significance 0.01 (bonferroni correction)
Statistical Analysis 2: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 1; Test type: Superiority; p = 0.376, Chi-squared, Corrected
Statistical Analysis 3: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 2; Test type: Superiority; p = 0.590, Chi-squared, Corrected
Statistical Analysis 4: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 3; Test type: Superiority; p = 0.320, Chi-squared, Corrected
Statistical Analysis 5: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 4; Test type: Superiority; p = 0.666, Chi-squared, Corrected

8. Secondary Outcome: Number of Patients With Sleep Problems
Description: Self-reported quality of sleep (days 0-4). Questionnaire. Results dichotomized to sleep problems (trouble falling asleep, frequent awakenings, no sleep) or no sleep problems.
Time Frame: 4 days
Population: Missing data from questionnaires, missing at random, not filled out or not sent back
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 26 | 25
Participants
  Day 0 | 13 | 12
  Day 1: number analyzed (Participants) | 25 | 23
  Day 1 | 9 | 13
  Day 2: number analyzed (Participants) | 25 | 22
  Day 2 | 8 | 9
  Day 3: number analyzed (Participants) | 23 | 20
  Day 3 | 9 | 9
  Day 4: number analyzed (Participants) | 22 | 19
  Day 4 | 8 | 8
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 0; Test type: Superiority; p > 0.999, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 1; Test type: Superiority; p = 0.154, Chi-squared, Corrected
Statistical Analysis 3: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 2; Test type: Superiority; p = 0.447, Chi-squared, Corrected
Statistical Analysis 4: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 3; Test type: Superiority; p = 0.678, Chi-squared, Corrected
Statistical Analysis 5: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 4; Test type: Superiority; p = 0.604, Chi-squared, Corrected

9. Secondary Outcome: Number of Patients With Feelings of Anxiety, Unrest and/or Sadness
Description: Self-reported feelings of anxiety, unrest, sadness (days 0-4). Questionnaire
Time Frame: postoperative day 0 to 4, once a day
Population: Missing data from questionnaires, missing at random
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 26 | 25
Participants
  Day 0 : sadness | 8 | 2
  Day 0 : restlessness | 11 | 8
  Day 0 : fatigue | 23 | 21
  Day 1 : sadness: number analyzed (Participants) | 25 | 23
  Day 1 : sadness | 6 | 4
  Day 1 : restlessness | 3 | 8
  Day 1 : fatigue | 20 | 17
  Day 2 : sadness: number analyzed (Participants) | 25 | 22
  Day 2 : sadness | 8 | 8
  Day 2 : restlessness | 6 | 11
  Day 2 : fatigue | 21 | 14
  Day 3 : sadness: number analyzed (Participants) | 23 | 20
  Day 3 : sadness | 9 | 6
  Day 3 : restlessness | 9 | 8
  Day 3 : fatigue | 17 | 13
  Day 4 : sadness: number analyzed (Participants) | 22 | 19
  Day 4 : sadness | 8 | 5
  Day 4 : restlessness | 10 | 3
  Day 4 : fatigue | 17 | 10
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 0, sadness; Test type: Superiority; p = 0.075, Chi-squared, Corrected
Statistical Analysis 2: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 0, restlessness; Test type: Superiority; p = 0.447, Chi-squared, Corrected
Statistical Analysis 3: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 0, fatigue; Test type: Superiority; p = 0.703, Chi-squared, Corrected
Statistical Analysis 4: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 1, sadness; Test type: Superiority; p = 0.731, Chi-squared, Corrected
Statistical Analysis 5: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 1, restlessness; Test type: Superiority; p = 0.052, Chi-squared, Corrected
Statistical Analysis 6: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 1, fatigue; Test type: Superiority; p = 0.807, Chi-squared, Corrected
Statistical Analysis 7: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 2, sadness; Test type: Superiority; p = 0.371, Chi-squared, Corrected
Statistical Analysis 8: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 2, restlessness; Test type: Superiority; p = 0.064, Chi-squared, Corrected
Statistical Analysis 9: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; day 2, fatigue; Test type: Superiority; p = 0.110, Chi-squared, Corrected
Statistical Analysis 10: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 3, sadness; Test type: Superiority; p = 0.531, Chi-squared, Corrected
Statistical Analysis 11: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 3, restlessness; Test type: Superiority; p = 0.954, Chi-squared, Corrected
Statistical Analysis 12: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 3, fatigue; Test type: Superiority; p = 0.526, Chi-squared, Corrected
Statistical Analysis 13: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 4, sadness; Test type: Superiority; p = 0.491, Chi-squared, Corrected
Statistical Analysis 14: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 4, restlessness; Test type: Superiority; p = 0.042, Chi-squared, Corrected
Statistical Analysis 15: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Day 4, fatigue; Test type: Superiority; p = 0.097, Chi-squared, Corrected

10. Secondary Outcome: Number of Patients Readmitted to Hospital Within 30 Days
Description: Any readmission within 30 days
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 32 | 32
Participants | 1 | 3
Statistical Analysis 1: Comparison: Dexamethasone 48 mg vs Dexamethasone 8 mg; Test type: Superiority; p = 0.613, Chi-squared, Corrected

11. Secondary Outcome: Number of Patients With Wound Infections Within 30 Days
Description: Any wound infections/complications
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
Number analyzed (Participants) | 32 | 32
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 hours after administration of trial drug(collection of possible adverse drug reactions), for readmissions and woundinfections: 30 days.
Arm/Group | Dexamethasone 48 mg | Dexamethasone 8 mg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone 48 mg (N=32) | Dexamethasone 8 mg (N=32)
bleeding, intraoperative (Surgical and medical procedures) | 1 (1) | 0 (0) — intraoperative bleeding, arterial damage

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT03161938/SAP_000.pdf
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT03161938/Prot_001.pdf